CLINICAL TRIAL: NCT04641702
Title: Comprehensive Assessment of Histopathologic and Physiologic Profile in Esophageal Motility Disorders
Brief Title: Comprehensive Esophageal Diagnostics Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anand Jain, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001665; 1K23DK131317-01A1 (NIH); 2025P013181 (Other: Emory IRB)
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Achalasia
Keywords: lower esophageal sphincter; Functional Lumen Imaging Probe Topography; anti-fibrosis agents; anti-inflammatory agents
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Intervention Model Description: Patients will have the option of consenting for Aim 1(pharmacologic challenge ), Aim 2 (in the event they go for future myotomy) or both if they choose to be included in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacologic challenge (Experimental): Measurement of esophageal response to atropine using functional lumen imaging probe (FLIP)
  Interventions: Drug: Atropine challenge; Procedure: Esophageal muscle biopsy

INTERVENTIONS:
Drug: Atropine challenge — Atropine challenge. After baseline FLIP, subjects will be administered 15 mcg/kg of intravenous atropine. Two minutes after administration, FLIP will be repeated.
Procedure: Esophageal muscle biopsy — Esophageal muscle biopsy. During standard-of-care Heller myotomy or per-oral endoscopic myotomy, 5mm of lower esophageal sphincter and distal esophageal circular muscle will be collected via biopsy forceps.

SUMMARY:
The prospective clinical trial will study muscle fibrosis in relation to lower esophageal sphincter (LES) measurements on Functional Lumen Imaging Probe (FLIP) Topography (the novel technology that utilizes impedance planimetry) after pharmacologic challenge. A better understanding of achalasia will allow intervention at an earlier stage.

DETAILED DESCRIPTION:
Achalasia is a disease characterized by inadequate opening of the lower esophageal sphincter. Achalasia is presumed to be due to neuronal dysfunction (active), however there are other variables such as muscle layer fibrosis (passive) that may contribute, particularly in milder or earlier achalasia variants. A new technology, impedance planimetry, may be able to measure active vs passive features of the lower esophageal sphincter (LES).

The prospective clinical trial will study muscle fibrosis in relation to lower esophageal sphincter (LES) measurements on Functional Lumen Imaging Probe (FLIP) Topography (the novel technology that utilizes impedance planimetry) after pharmacologic challenge. A better understanding of achalasia will allow intervention at an earlier stage.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age 18 and above.
2. Evaluated by Emory Digestive Diseases Clinic, Emory Motility Lab, the Emory Endoscopy Unit, or Emory Surgery Department starting October 1, 2020.
3. Has a diagnosis of achalasia or an esophageal motility disorder with confirmed evaluation by one of the following modalities: functional lumen imaging probe (FLIP) or high-resolution esophageal manometry (for Aim 1)
4. Undergoing a diagnostic Functional Lumen Imaging Probe (FLIP) study at Emory University Hospital with anesthesia assistance (for Aim 1)
5. Undergoing Heller myotomy or per oral endoscopic myotomy for the treatment of their esophageal motility disorder (for Aim 2)

Exclusion Criteria:

1. Patients younger than 18 years old
2. Pregnant women
3. Prisoners
4. Non-English speaking - the rationale is that the symptom characterization and outcome data are measured on detailed and fairly lengthy (5-7 pages) questionnaires written in English with some medical terms. These are standardized questionnaires with no short forms available.
5. Cognitively impaired adults unable to provide informed consent
6. Cardiac disease in the form of - arrhythmia requiring ICD or pacemaker, baseline bradycardia with HR <60 or tachycardia with HR > 90, congestive heart failure with ejection fraction <35%, history of myocardial infarction, baseline MAP <65 or systolic BP >140, asthma or chronic obstructive pulmonary disease, urinary retention requiring the use of foley catheterization (including intermittent use), narrow-angle glaucoma, myasthenia gravis, GFR <60 [exclusions for Aim 1 only]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of lower esophageal sphincter contraction and relaxation | Two minutes after the study drugs administration
  Degree of lower esophageal sphincter contraction and relaxation will be measured
The collagen content in muscle biopsy specimens | Two minutes after the study drugs administration
  The collagen content in muscle biopsy specimens will be measured on Sirius Red and Masson Trichrome staining.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Jain, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Esophageal function testing data, symptom questionnaire data, treatments performed, and biospecimen analysis results will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Estimated January 2025.
Access Criteria: Collaborators with whom the study team has Data Use Agreements in Place will have access through secure electronic means.